CLINICAL TRIAL: NCT04409470
Title: Venous Versus Arterial Blood Gas Sampling in Undifferentiated Emergency Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, PhD, Emergency department head of research, University Hospital, Linkoeping
Other Study IDs: SE2020-00396
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Dyspnea; Hypercapnia
Keywords: arterial blood gas; venous blood gas
MeSH Terms: conditions — Dyspnea; Hypercapnia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood from arterial and venous puncture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indication for blood gas sampling: To be eligible, patients will need to be classified as critically ill and there has to be a clear clinical indication for an arterial blood gas sampling. Enrollment will be performed in a consecutive manner at all hours.
  Interventions: Diagnostic Test: Blood gas sampling from artery and vein

INTERVENTIONS:
Diagnostic Test: Blood gas sampling from artery and vein — Patients included in this study are treated according to clinical routine. After inclusion, sampling of an arterial blood gas and a venous blood gas is performed simultaneously or as close in time as possible. Because the venous blood gas analysis sample can be taken directly from the patient's peripheral venous catheter, no additional venous puncture is usually required and the additional amount of blood that may be required is approx. 1 ml (the assay requires about 500 µl). In the very rare cases where it is not possible to establish a peripheral venous catheter within a reasonable time, the sample will be acquired from a new venous puncture together with other venous routine samples.

SUMMARY:
In the emergency department and intensive care unit, blood gas analysis is a crucial tool in the assessment of critically ill patients. Blood gas analysis is quick and repeatable at the bedside. The sampling can be done from both arterial and venous samples, with arterial samples generally considered to be more reliable and by that widely used as the standard method.

The purpose of this project is to compare venous and arterial blood gas parameters in undifferentiated, critically ill patients. We plan to evaluate the correlation between different parameters through a prospective observational study. In particular, carbon dioxide partial pressure (pCO2) correlation between venous and arterial samples is investigated by using and comparing different conversion models proposed in the literature.

250 patients deemed to be in need of arterial blood gas sampling based on their clinical condition will be included in a consecutive fashion at all hours.

The long-term goal is to clinically translate the findings into a limitation on the use of arterial sampling, which could potentially reduce pain and complication risks in the many patients who undergo arterial blood gas sampling every day.

DETAILED DESCRIPTION:
== Practical procedures & flowchart ==

Patients included in this study are treated according to clinical routine. After inclusion, sampling of an arterial blood gas and a venous blood gas is performed simultaneously or as close in time as possible. Because the venous blood gas analysis sample can be taken directly from the patient's peripheral venous catheter, no additional venous puncture is usually required and the additional amount of blood that may be required is approx. 1 ml (the assay requires about 500 µl). In the very rare cases where it is not possible to establish a peripheral venous catheter within a reasonable time, the sample will be acquired from a new venous puncture together with other venous routine samples.

Sampling can be carried out by doctors or nurses. The arterial and venous blood gas analysis is performed with a blood gas analyzer (ABL90) in the emergency department and is performed immediately after the sampling. Sampling times and analysis times are documented.

Survey results are routinely stored in electronic form in patient health record and also locally on the device ABL90 with social security number as ID. The data is saved for statistical analysis.

== Documentation ==

The following parameters are documented during sampling:

* Chief complaint
* Indication for sampling
* The patient's current vital signs at the time of sampling
* Ongoing oxygen treatment (flow rate)
* Size of cannula, sampling location
* Sampling times and analysis times
* Number of puncture attempts

After sampling, the following is documented:

* Analysis results of venous and arterial blood gas sample
* Final diagnosis at discharge from the emergency department

The documentation will primarily be on worksheets, which will be marked with a patient label (name / social security number) and a serial number. The worksheet will be stored together with consent forms in a locked space of Akutkliniken US Linköping.

The data will be archived in the local emergency department or at the Regional Archives in Östergötland according to applicable laws and regulations.

The result of blood gas analysis is obtained from the digital lab system in the patient record (Lab-ROS) or directly exported from the internal memory of the analyzers at the emergency department. In both cases, the results will be used for digital compilation of study data. All electronic storage of study data will be pseudonymized by linking to patients serial number.

== Statistics ==

In previous studies, the correlation between arterial and venous samples has been evaluated using several different statistical methods:

* T-test, Pearson's and Spearman's R variable
* Descriptive data are presented as mean and +/- from SD

Our intention in this study is to make a parallel comparison of previously published methods, as well as to examine, based on collected data, whether a new formula with better precision can be derived.

== The potential significance of the project ==

At present, arterial blood gas sampling is used as the standard procedure for assessing a critically ill patient in the emergency department.

The project aims to clarify the feasibility of replacing routine arterial blood gas sampling in the emergency department with venous punctures without impairing test results and patient care. If feasible, such a change in sampling routines could potentially mean a great improvement for patients in terms of pain and complication risks. Also, workflow and lead times in the emergency department could be improved by the fact that venous samples may be drawn by all clinical staff, whereas arterial samples are normally reserved for doctors and nurses with dedicated training.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to understand and process oral and written information and give his/her consent (within 12h), or consent provided by a close relative.
* Aged > 18 years
* Assessed to be in need of arterial blood gas analysis

Exclusion Criteria:

* Unwilling to participate, or unable to understand the provided information
* Inability to give subsequently consent (> 12 hours) or unwillingness by close relative to provide consent.
* Pregnant
* Aged < 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For enrolment, we will consider all patients who are admitted to the emergency department irrespective of mode of arrival (ambulance, walk-in etc). To be eligible, patients will need to be classified as critical ill and there has to be a clear clinical indication for an arterial blood gas sampling. Indications for arterial blood gas sampling, in turn, are primarily dictated by local SOPs (Standard Operating Procedures; "PM/ vårdprocessåtgärder") for appropriate sampling based on chief complaint, age, and vital signs upon arrival. The aim is to include these patients consecutively around-the-clock.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-03-27 (Actual)

PRIMARY OUTCOMES:
How does pCO2 correlate between arterial and venous blood gas samples? | October - November 2020
Can a clinically reliable correlation be identified using a conversion model? (existing or new) | October - November 2020

SECONDARY OUTCOMES:
How does processing times and sampling location affect the result? | October - November 2020
How does the patient's vital parameters (blood pressure, pulse) affect the results? | October - November 2020
In there a difference in the analysis results between the emergency department and the central laboratory? | October - November 2020
How reliable are the results beyond mild to moderate deviations from normal values in consecutive enrolled, critically ill patients? | October - November 2020

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Jörg, MD, Principal Investigator — Emergency Department, University Hospital Linköping, Sweden
Locations (1):
- University Hospital Linköping, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bengezi OA, Dalcin A, Al-Thani H, Bain JR. Unusual complication of radial artery cannulation. Can J Plast Surg. 2003 Winter;11(4):213-5. doi: 10.1177/229255030301100409. PMID 24009442
- [Background] Bloom BM, Grundlingh J, Bestwick JP, Harris T. The role of venous blood gas in the emergency department: a systematic review and meta-analysis. Eur J Emerg Med. 2014 Apr;21(2):81-8. doi: 10.1097/MEJ.0b013e32836437cf. PMID 23903783
- [Background] EMCrit, About, Josh Farkas, and The Emcrit Crew. 2017. "PulmCrit- How to Convert a VBG into an ABG." EMCrit Project. January 16, 2017. https://emcrit.org/pulmcrit/vbg-abg/.
- [Background] Giner J, Casan P, Belda J, Litvan H, Sanchis J. [Use of the anesthetic cream EMLA in arterial punction]. Rev Esp Anestesiol Reanim. 2000 Feb;47(2):63-6. Spanish. PMID 10769553
- [Background] Hess D, Agarwal NN. Variability of blood gases, pulse oximeter saturation, and end-tidal carbon dioxide pressure in stable, mechanically ventilated trauma patients. J Clin Monit. 1992 Apr;8(2):111-5. doi: 10.1007/BF01617428. PMID 1583545
- [Background] Jang JS, Jin HY, Seo JS, Yang TH, Kim DK, Kim DK, Kim DI, Cho KI, Kim BH, Park YH, Je HG, Kim DS. The transradial versus the transfemoral approach for primary percutaneous coronary intervention in patients with acute myocardial infarction: a systematic review and meta-analysis. EuroIntervention. 2012 Aug;8(4):501-10. doi: 10.4244/EIJV8I4A78. PMID 22581470
- [Background] Kelly AM, McAlpine R, Kyle E. How accurate are pulse oximeters in patients with acute exacerbations of chronic obstructive airways disease? Respir Med. 2001 May;95(5):336-40. doi: 10.1053/rmed.2001.1046. PMID 11392573
- [Background] Kelly AM. Can VBG analysis replace ABG analysis in emergency care? Emerg Med J. 2016 Feb;33(2):152-4. doi: 10.1136/emermed-2014-204326. Epub 2014 Dec 31. PMID 25552544
- [Background] Lemoel F, Govciyan S, El Omri M, Marquette CH, Levraut J. Improving the validity of peripheral venous blood gas analysis as an estimate of arterial blood gas by correcting the venous values with SvO(2). J Emerg Med. 2013 Mar;44(3):709-16. doi: 10.1016/j.jemermed.2012.07.041. Epub 2012 Aug 24. PMID 22921853
- [Background] Malatesha G, Singh NK, Bharija A, Rehani B, Goel A. Comparison of arterial and venous pH, bicarbonate, PCO2 and PO2 in initial emergency department assessment. Emerg Med J. 2007 Aug;24(8):569-71. doi: 10.1136/emj.2007.046979. PMID 17652681
- [Background] O'Connor TM, Barry PJ, Jahangir A, Finn C, Buckley BM, El-Gammal A. Comparison of arterial and venous blood gases and the effects of analysis delay and air contamination on arterial samples in patients with chronic obstructive pulmonary disease and healthy controls. Respiration. 2011;81(1):18-25. doi: 10.1159/000281879. Epub 2010 Feb 4. PMID 20134147
- [Background] Scheer B, Perel A, Pfeiffer UJ. Clinical review: complications and risk factors of peripheral arterial catheters used for haemodynamic monitoring in anaesthesia and intensive care medicine. Crit Care. 2002 Jun;6(3):199-204. doi: 10.1186/cc1489. Epub 2002 Apr 18. PMID 12133178
- [Background] Shah, Shobhit, and Department of Medicine and Pulmonology, Mata Chanan Devi Hospital, Janakpuri, New Delhi. 2017. "Comparison and Agreement between Venous and Arterial Blood Gas Values for pH, pCO2, pO2, Bicarbonate and Oxygen Saturation in Patients with Acute Respiratory Illnesses." Journal of Medical Science And Clinical Research 05 (03):19069-70.
- [Background] Shirani F, Salehi R, Naini AE, Azizkhani R, Gholamrezaei A. The effects of hypotension on differences between the results of simultaneous venous and arterial blood gas analysis. J Res Med Sci. 2011 Feb;16(2):188-94. PMID 22091230
- [Background] Thorson SH, Marini JJ, Pierson DJ, Hudson LD. Variability of arterial blood gas values in stable patients in the ICU. Chest. 1983 Jul;84(1):14-8. doi: 10.1378/chest.84.1.14. PMID 6407807
- [Background] Zeserson E, Goodgame B, Hess JD, Schultz K, Hoon C, Lamb K, Maheshwari V, Johnson S, Papas M, Reed J, Breyer M. Correlation of Venous Blood Gas and Pulse Oximetry With Arterial Blood Gas in the Undifferentiated Critically Ill Patient. J Intensive Care Med. 2018 Mar;33(3):176-181. doi: 10.1177/0885066616652597. Epub 2016 Jun 9. PMID 27283009
- See also: Complete study protocol as used for approval at the Swedish Ethical Review Authority — https://docs.google.com/document/d/1O2IORTvjj9ElWMuTgIIEONGvXUxefBRQ7-H5NQk9r8Q/edit?usp=sharing